CLINICAL TRIAL: NCT04019522
Title: An Exploration of Acute Intermittent Hypoxia as a Tool to Enhance Neural Recovery in Stroke Survivors; a Pilot Safety Study.
Brief Title: American Heart Association- Stroke/Hypoxia Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Zev Rymer, Director Single Motor Unit Laboratory, Research Arms + Hands Lab, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU: 00208610
Record Dates: First submitted 2019-06-19; First posted 2019-07-15 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoxia (Experimental): During each session, study participants will receive a single sequence of AIH, consisting of 15 x 60-seconds periods of hypoxia alternating with 90-seconds of normoxia (21% O2), for a total of 30 minutes, whilst in a seated upright position. AIH will be applied by directing gas flow to a reservoir bag connected via plastic tubing to a non re-breathing facemask/respiratory valve system while the participants are in a seated position. Defined gas mixtures will be delivered by manual adjustment of one-way valves attached to a hypoxia generator.
  Interventions: Other: Acute Intermittent Hypoxia (AIH)

INTERVENTIONS:
Other: Acute Intermittent Hypoxia (AIH) — An oxygen monitor will continuously measure and record the fraction of inspired oxygen delivered to the subject. Inspired fraction of oxygen (FiO2) of the gas mixture will be individually adjusted using the valve settings to reach the targeted SpO2. The gas mixtures administered during the four sessions will be 21% O2 (target SpO2 = 95%), 17% O2 (target SpO2 = 92%), 13% O2 (target SpO2 = 87%) and 9% O2 (target SpO2 = 82%).

SUMMARY:
Of the 795,000 people who experience a stroke every year in the US, only a small percentage will achieve full recovery. While current therapies promote strength and endurance, none directly address the unique potential of the brain to reorganize following injury. The goal of this project is to explore the effects of a novel therapy, acute intermittent hypoxia (AIH). During this therapy, individuals receive brief bouts of reduced oxygen levels by inhalation through a face mask. (This is akin to being on top of a tall mountain). In brief exposures, AIH is known to trigger the release of specific proteins that help the brain adapt to oxygen reductions. Published results in people with incomplete spinal cord injury have shown that AIH enhances muscle strength and coordination rather quickly. The research team aims to study the effects of AIH in stroke survivors.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death and a leading cause of long-term disability worldwide. Despite the spontaneous recovery that occurs following a hemispheric stroke, more than half of stroke patients show substantial residual impairments, imposing a significant human and economic burden. This burden is likely to increase in coming decades, due to a rapidly aging population, and the associated progression of cardiovascular risk factors. Accordingly, new interventions to alleviate impairment in stroke survivors are urgently needed. The development and testing of one such novel intervention, termed Acute Intermittent Hypoxia (AIH), is the primary focus of this AHA Innovative Project Award.

The aim is to answer questions related to safety and preliminary efficacy of AIH in stroke survivors. First, the Investigators will establish whether brief reductions in inhaled oxygen concentration can be safely tolerated in stroke survivors. A clinician will closely monitor subjects for any adverse events.

The second aim is to establish the effects of AIH on elbow flexion/extension strength, and on hand grip and pinch strength. Subjects will be monitored closely for any adverse events during these experiments. Data will be analyzed to determine if there is an improvement in key outcomes at any dose level.

ELIGIBILITY:
Inclusion criteria:

Age ≥18 years;

A first time, unilateral, ischemic, hemispheric stroke, confirmed by magnetic resonance imaging (MRI);

Chedoke assessment > 3

Ability to open and close affected hand

Able to understand and communicate in English

Be able to consent independently

≥ 6 months post stroke

Must have a hemoglobin level above 10g/dl (to be confirmed using handheld noninvasive lab equipment)

Must have ability to attend research visits with a companion for assistance

WOCBP must be comfortable confirming negative pregnancy prior to hypoxia experimental therapy.

Exclusion criteria:

Brain stem or cerebellar stroke; mean Fazekas score rated on initial fluid-attenuated inversion recovery MRI ≥3

Severe aphasia, preventing subject from understanding the protocol and giving written consent;

History of prior neurological disorder;

Pre-existing hypoxic pulmonary disease,

Severe hypertension (>160/100)

Ischemic cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical/neurological status over the duration of the study | 6 days
  All adverse events will be reviewed for safety and study continuation by the medical monitor.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | 6 days
  is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score ranging from 0-42.
Fugl- Meyer Assessment | 6 days
  Each test element will be graded on a 3-point ordinal scale and summed up to provide a maximum upper limb score of 66. Reliability and validity have been demonstrated. The FMA will be administered while the subject is seated.
Modified Ashworth Scale | 6 days
  This scale allows for characterization of increases in muscle tone, from low or normal tone to complete limb rigidity. Specifically, we will evaluate the elbow flexors, bilaterally
Grip strength | 6 days
  A dynamometer measures maximum gross grasp (lb.) averaged over three attempts with each hand. The minimum possible value of zero lb. will be assigned when the participant cannot actively flex the fingers or grasp the dynamometer. Completed bilaterally, if possible
Pinch Strength | 6 days
  Hydraulic Handheld Dynamometer): A dynamometer measures maximum gross grasp (lb.) averaged over 3 attempts with each hand. The minimum possible value of zero lb. will be assigned when the participant cannot actively flex the fingers or grasp the dynamometer.
Elbow strength | 6 days
  monitoring changes in isometric elbow flexion force using a dynamometer. A total of three trials will be taken on each side, with a rest break between trials. The average of the three trials will be recorded.
D-KEFS Color-Word Interference Test | 6 days
  A neuropsychological measure that seeks to evaluate attention and inhibition. Subjects will be asked to read words or name ink colors as quickly as possible within a given time limit. The test supplies the examiner with three separate scores, including an ability to calculate an interference score. This final score allows for interpretation of cognitive flexibility, creativity and cognitive stress. This measure will be utilized to monitor subjects throughout their participation at specific time-points. Audio recording may be taken to ensure accurate recording of responses
5 minute neurological test | 6 days
  Quick short tests to assess clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Zev Rymer, MD/PhD, Principal Investigator — Principal Investigator
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pearcey GEP, Barry AJ, Sandhu MS, Carroll TJ, Roth EJ, Rymer WZ. Acute Intermittent Hypoxia in People Living With Chronic Stroke: A Case Series. Stroke. 2025 Apr;56(4):1054-1057. doi: 10.1161/STROKEAHA.124.046620. Epub 2025 Feb 25. PMID 39996325